CLINICAL TRIAL: NCT06861387
Title: A Randomized Controlled Trial Studying the Effect of Additional Intercostal Cryo-analgesia (ICCA) to Standard Postoperative Pain Management in Patients Undergoing Minimally Invasive Lung Surgery
Brief Title: Cryo Nerve Block Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, B.T.G. Köhlen, Coordinating investigator, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL88359.100.24
Record Dates: First submitted 2024-11-18; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-11

CONDITIONS: Intercostal Nerve Block; Cryo Analgesia; Minimally Invasive Lung Surgery
Keywords: cryo analgesia; intercostal nerve block; minimally invasive lung surgery; pain management
MeSH Terms: conditions — Agnosia | interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: Single centre, blinded randomized controlled
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cryo-analgesia (Experimental): The intervention group will receive intercostal cryo-analgesia and standard postoperative pain management including intercostal nerve block, patient conrolled analgesia, and acetaminophen.
  Interventions: Device: Cryotherapy; Drug: PAiN - multimodal analgesia
- Standard care (Active Comparator): The control group will receive standard postoperative pain management including intercostal nerve block, patient conrolled analgesia, and acetaminophen.
  Interventions: Drug: PAiN - multimodal analgesia
- Registry (Other): The registry group will receive intercostal cryo-analgesia and standard postoperative pain management including intercostal nerve block, patient conrolled analgesia, and acetaminophen. Patient are eligible for the registry group in case they refuse randomization
  Interventions: Device: Cryotherapy; Drug: PAiN - multimodal analgesia

INTERVENTIONS:
Device: Cryotherapy — AtriCure's cryoICE cryoSPHERE probe will be inserted through one of the incisions used for VATS/RATS. Cryo-analgesia will be performed unilaterally on the intercostal nerve at the level Th3-Th7. Thus, cryo-analgesia will be applied on 5 intercostal levels. The probe will be placed at the inferior aspect of the ribs, posterior to the mid-axillary line, directly on the neurovascular bundle. One freezing cycle takes approximately 2 minutes and a temperature of between minus 50 and 70 degrees Celsius will be applied.
  Arms: Cryo-analgesia; Registry
Drug: PAiN - multimodal analgesia — Our standard postoperative pain management plan consists of intercostal nerve block, patient controlled analgesia and acetaminophen

SUMMARY:
Background Minimally invasive lung surgery, such as video-assisted thoracoscopic surgery (VATS) or robot-assisted thoracoscopic surgery (RATS), has become more common for lung resections because it leads to faster recovery, less pain, and shorter hospital stays. However, pain after surgery remains a major issue. Current guidelines suggest using a combination of pain management strategies to reduce the use of opioids and their side effects. Intercostal cryo-analgesia (ICCA), a technique that uses cold to reduce nerve activity, may help lower pain and opioid use after surgery. However, there is limited research on ICCA, with most studies having small sample sizes and lacking randomized controlled trials. More research is needed to compare ICCA with standard pain management in patients having minimally invasive lung surgery.

Objective:

The goal of this study is to determine if ICCA improves recovery compared to the standard pain management after minimally invasive lung surgery. We aim to measure recovery time and quality using the Quality of Recovery 15 (QoR-15) questionnaire. We expect that ICCA will result in better recovery, less pain, less use of opioids, and shorter hospital stays, without increasing the risk of nerve damage or other complications.

Study Design:

This will be a single-center, blinded, randomized controlled trial, along with an observational registry.

Study Population:

The study will include adults who are having elective minimally invasive lung resections.

Intervention:

Patients in the intervention group will receive ICCA in addition to the standard pain management after surgery. ICCA will be administered by the surgeon before closing the wound, targeting the intercostal nerves between ribs 3 and 7.

Main Study Parameters/Endpoints:

The main outcome will be recovery time, measured using the QoR-15 questionnaire. The QoR-15 assesses overall recovery after surgery across several areas, with a score of 118 or higher indicating good recovery. The questionnaire is a reliable and valid tool to measure recovery from surgery.

Risks and Benefits:

This trial will examine the effects of adding ICCA to the standard pain management protocol. Potential risks include numbness or nerve damage, neuropathic pain (pain caused by nerve injury), or complications like bleeding (hematoma) or lung collapse (pneumothorax) at the treatment site. The potential benefits of ICCA include better recovery, reduced opioid use, less pain, shorter hospital stays, and fewer breathing problems after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are at least 18 years or older.
2. Patients are electively scheduled to undergo minimally invasive (i.e., VATS or RATS) anatomical lung (i.e., pneumonectomy, (bi)lobectomy, or segmentectomy) resection for benign or malignant disease.
3. Proficient understanding of the consequences of enrolment by the patients.
4. Written informed consent by the patient.

Exclusion Criteria:

1. Patients with reported intolerance or hypersensitivity to the anaesthetic drug used for ICNB.
2. Patients chronically using opioids for reasons not related to the operation (i.e., more than 3 months).
3. Patients with liver failure inhibiting the systematic use of acetaminophen (i.e., paracetamol)
4. Patients with connective tissue disease.
5. Patients with comorbidities or history contra-indicating ICCA.
6. Patients who are pregnant.
7. Participation in other clinical trial(s) that may interfere with the current trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-12 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery | 6 months
  Quality of Recovery based on the Quality of Recovery (QoR-15) questionnaire, whereas a minimum of 118 points correspondents with a clinically good recovery

SECONDARY OUTCOMES:
Pain scores | 6 months
  In-hospital and outpatient pain scores are based on the numeric rating scale (NRS), whereas score 0 means "no pain" and 10 "extreme pain"
Postoperative opioid consumption | 6 months
  In-hospital and outpatient postoperative opioid consumption is measured in MME use.
Concomittant analgesia | 6 months
  use of concomittant analgesia
Postoperative complications | 6 months
  1. Surgery-related complications.
  2. Surgical site infection.
  3. Respiratory tract infections/pneumonia.
  4. Pneumothorax.
  5. Chest wall hematoma.
Length of stay hospital | 6 months
  Length of stay hospital
Operative time | 6 months
  Total operative time

OTHER OUTCOMES:
Presence of neuropathic pain or other sensory changes | 6 months
  hypesthesia, hyperesthesia and/or allodynia
Prolonged analgesia | 6 months
  Prolonged analgesia more than 3 months after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- St. Antonius Ziekenhuis, Nieuwegein, Utrecht, Netherlands